CLINICAL TRIAL: NCT01495286
Title: Is the Use of Noninvasive Electrical Stimulation of Acupuncture Points (NESAP) During a Routine Heelstick Safe in Infants?
Brief Title: Safety of Noninvasive Electrical Stimulation of Acupuncture Points (NESAP) in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114283
Record Dates: First submitted 2011-12-09; First posted 2011-12-20 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-10

CONDITIONS: Pain
Keywords: newborn infant; acupuncture; safety; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: EMPI Select Transcutaneous Electrical Nerve Stimulation — Experimental: EMPI Select TENS unit For analgesia, StimCare electrodes will be placed on the baby's legs at specific acupuncture points and electrical stimulation will be administered via a standard EMPI Select TENS unit. For the main study, a low continuous current will be provided with voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 5±1 min after the heel stick. Two sub studies will precede the main safety study, with 6 infants in each, using electrical stimulation intensities that are a fraction of the planned intensity. Infants in sub study 1 will receive electrical stimulation at 1 mA and 2 Hz. Infants in sub study 2 will receive electrical stimulation at 2 mA and 10 Hz.
  Other Names: Noninvasive electrical stimulation

SUMMARY:
This research study represents a pilot, open arm study that will evaluate the safety of using Non-invasive Electrical Stimulation of Acupuncture Points (NESAP) in 42 newborn infants less than 3 days of age who require heel sticks for clinical blood sampling. The investigators plan to enroll 51 infants into the study in order to obtain 42 completed infants. Two sub studies will precede the main safety study, with 6 infants in each sub study and 30 infants in the main study. These two sub studies will use electrical stimulation intensities that are a fraction of the planned intensity of electrical stimulation that will be used during the main part of the study.

The clinical trial will be performed at the University of Arkansas for Medical Sciences Hospital (Little Rock, AR). The study will evaluate the pain response to heel stick routinely used to obtain This blood from 30 term neonatal infants, ages 37 to 42 weeks Electrical stimulation will be applied at appropriate acupuncture points using a very low current for 10 minutes, routine for procedural pain. The response to pain will be assessed using pain scales and physiologic changes.

The investigators hypothesize that the NESAP procedure is safe in newborn infants undergoing a routine heelstick.

DETAILED DESCRIPTION:
The investigators propose an open label trial to assess the safety of using electrical stimulation at acupuncture sites in 42 infants receiving a routine heel stick. Two sub studies will precede the main safety study, with 6 infants in each sub study and 30 infants in the main study. These sub studies will use electrical stimulation intensities that are a fraction of the planned intensity of the electrical stimulation that will be used for the main part of the study.

As part of routine neonatal screening, blood will be collected from a heel stick(s) by qualified nursing staff in the hospital nursery or in the patient's room. Less than one ml of blood will be drawn over 1-2 minutes. Study infants will be watched more carefully with heart rate, respiratory rate, and oxygen saturation performed as part of this study. Infants not participating in the study will be watched as per usual unit protocol.

Electrical stimulation at acupuncture sites will be administered via an EMPI Select Transcutaneous Electrical Nerve Stimulation (TENS) unit. To produce analgesia, small electrodes will be placed on the baby's legs at specific acupuncture points: ZuSanLi (ST36) just below the knee, triggers release of endorphins; SanYinJiao (SP6) just above the inner ankle, important point for energy balance; Kun Lun (BL60) depression behind lateral malleolus, protects local tissue trauma to heel; and Tai Xi (Ki3) behind the inner ankle, an important energy meridian. 25, 39, 48-50, StimCare self-adhesive electrodes with a gel base will be applied to the skin; the skin will not be punctured by these procedures. For the main part of the study, a low continuous current will be provided with minimal voltage of 3.5 milliamps (mA). The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 5±1 min after the heelstick. This paradigm is based on the basic animal research developed by Dr. Han and other research groups. Two sub studies will precede the main safety study, with 6 infants in each sub study, using electrical stimulation intensities that are a fraction of the planned intensity. Infants in sub study 1 will receive electrical stimulation at 1 mA and 2 Hz. Infants in sub study 2 will receive electrical stimulation at 2 mA and 10 Hz.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants born at 37-42 weeks gestational age and less than 3 days of age requiring a heelstick for clinically indicated blood sampling.
* A normal neurological assessment

Exclusion Criteria:

* Newborns who have received any analgesic treatment
* Infants exposed to chronic opiates in utero (excluding opiates given only at the time of delivery) or with a positive drug screen based on review of medical records
* Infants exposed to birth asphyxia (5-minute Apgar scores of <5 or cord pH <7.0).
* Infants on mechanical ventilation.
* Newborns with suspected or confirmed neuromuscular diseases, congenital anomalies, or sepsis.
* Infants with birth trauma to the lower extremities (bruising or other) or those exposed multiple heelsticks in the previous 24 hours (e.g. requiring frequent glucose or bilirubin measurements).
* Infants born from mothers with drug addiction, diabetes, pre-eclampsia, or systemic inflammatory conditions.
* Infants with abnormal neurological exams
* Infants with congenital heart defects
* Any condition the investigator determines will put the subject at risk if participating in the study.
* Enrollment / participation in other studies
* Dermatological condition(s) in the area of electrode placement or elsewhere
* Local or systemic infection documented or suspected
* Allergy to the gel or adhesive
* Bleeding abnormalities
* Connection to other medical equipment or devices that may interfere with the workings or functioning of the TENS unit

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hall, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period started 12/15/11, ended 06/21/12. All recruitment took place in the well mothers and babies (rooming-in) unit at the University of Arkansas Medical Center (UAMS). Parents of infants were contacted in their individual rooms by research staff and parents signed IRB -approved consents if they wanted their infants to participate.
Pre-assignment Details: The parents of one infant signed the consent form but then changed their minds before the infant actually participated in the study. This infant was withdrawn from the study.
Groups:
- Noninvasive Electrical Stimulation Acupuncture Points (NESAP): This was a single arm study, a descriptive pilot study to assess the safety of using noninvasive electrical stimulation at acupuncture points (NESAP) as an analgesic during routine heel sticks for newborn screenings. All infants who participated in the study received NESAP starting 10 minutes before the heel stick. The treatment continued throughout the heel stick and for 5 minutes afterwards. The first 6 infants received NESAP with an Empi Select transcutaneous electrical nerve stimulation (TENS) unit at 1.0 mA, 2 Hz. THe second 6 infants received TENS unit stimulation at 2.0 mA, 10 Hz. The last 18 infants received TENS unit stimulation at 3.5 mA, 10 Hz.
Period: Overall Study
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: days] | 1 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate During Treatment With TENS Unit
Description: Changes in heart rate will be recorded after an initial baseline heart rate. Heart rate will be taken at baseline, after 5 minutes of NESAP, at 5 minutes after end of heel stick, and upon return to infant's room.
Time Frame: Duration of the TENS unit treatment and heel stick, an expected average of 20 minutes.
Population: We based power analysis on 90% power for detecting that the PIPP score had increased by 4, indicating a significant change. With 30 infants, we had 90% power for detecting whether the pain score (PIPP) had increased significantly when testing with a .05 level, one-sided paired t-test.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Number analyzed (Participants) | 30
beats per minute
  Baseline heart rate | 137 (11.9)
  Heart rate after 5 minutes of NESAP | 131 (15)
  Heart rate 5 minutes after heelstick | 133 (15)
  Heart rate after return to room | 133 (15)

2. Primary Outcome: Oxygen Saturation During Treatment With TENS Unit and Routine Heel Stick
Description: Changes in oxygen saturation after an initial baseline oxygen saturation. Oxygen saturation will be measured after TENS unit is initiated, for 10 minutes between TENS initiation and heel stick,during heel stick, and for 5 minutes afterwards. Measurements will be taken at baseline, after 5 minutes of NESAP, and at 5 minutes after end of heel stick.
Time Frame: Baseline, duration of the TENS unit treatment and heel stick, an expected average of 20 minutes.
Population: We based power analysis on 90% power for detecting that the PIPP score had increased by 4, indicating a significant increase in pain level. With 30 infants, we had 90% power to detect a significant increase in PIPP score with a .05 level, one-sided paired t-test.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Number analyzed (Participants) | 30
percentage of oxygen saturation
  Oxygen saturation before NESAP | 98 (1.55)
  Oxygen saturation after 5 minutes of NESAP | 97 (2.18)
  Oxygen saturation 5 minutes after heel stick | 96 (2.3)

3. Secondary Outcome: Blood Pressure During TENS Treatment and Heel Stick
Description: Changes in systolic and diastolic blood pressure after initial baseline. Measurements will be taken at baseline, after 5 minutes of NESAP, at 5 minutes after end of heel stick, and upon return to infant's room.
Time Frame: Duration of the TENS unit treatment and heel stick, an expected average of 20 minutes.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Number analyzed (Participants) | 30
mm Hg
  Systolic blood pressure before NESAP | 85 (13)
  Systolic blood pressure after 5 minutes NESAP | 84 (12)
  Systolic blood pressure 5 minutes after heel stick | 84 (13)
  Systolic blood pressure after return to room | 83 (10)

4. Secondary Outcome: Pain During TENS Treatment and Routine Heel Stick
Description: Pain scores were measured using the Premature Infant Pain Profile (PIPP). The PIPP is a composite pain tool that measures pain based on behavioral and physiologic parameters and adjusts for gestational age. Differences in pain scores were recorded throughout the heel stick process, using a baseline score as reference. Mean pain scores were calculated before NESAP (baseline), after the TENS unit was turned on, after ten minutes of NESAP but before heel stick, during heel cleaning, during the initial heel stick, during heel squeeze, and during recovery. For term infants, the range of PIPP scores is on a scale of 0 for no pain to 18 for severe pain. A score of 6 indicate mild pain, and a score of 11 -12 indicates moderate pain. An increase in PIPP score of 4 or greater from baseline indicates a significant change in pain level.
Time Frame: Pain score given during the heel stick process and for 2 minutes afterwards
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Number analyzed (Participants) | 30
units on a scale
  Pain score (PIPP) before NESAP | 2.17 (1.72)
  Pain score (PIPP) after TENS unit turned on | 2.8 (2.14)
  Pain score (PIPP) after 10 minutes of NESAP | 1.57 (1.3)
  Pain score (PIPP) during heel cleaning | 3.17 (2.09)
  Pain score (PIPP) during heel stick | 8.88 (4.26)
  Pain score (PIPP) during heel squeeze | 8.13 (4.2)
  Pain score (PIPP) during recovery | 4.32 (3.76)

5. Secondary Outcome: Skin Assessment
Description: Areas of skin where the Stim Care electrodes are placed will be assessed for redness, tenderness, or any other change in skin condition. Assessment will take place at baseline, after the NESAP procedure, upon discharge from the hospital, and after one week. If there is a problem at one week, there will be additional follow-up at two weeks.
Time Frame: Post procedure monitoring for the duration of the hospital stay, an expected average of 1 day. Follow up phone calls at one week and again at two weeks if needed.
Population: We based power analysis on 90% power for detecting that the PIPP score had increased by 4, indicating a significant change. With 30 infants,we had 90% power for detecting whether the pain score (PIPP) had increased significantly when testing with a .05 level, one sided paired t test
Measure: Number; unit: participants
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Number analyzed (Participants) | 30
participants
  Baseline assessment for skin irritation | 0
  Skin irritation after NESAP | 0
  Skin irritation upon discharge | 0
  Skin irritation after one week | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Monitored before, during, and after NESAP for heart rate, oxygen saturation, blood pressure, seizure activity, emesis, color change, skin changes, muscle tone changes. One week follow-up by phone.
Arm/Group | Noninvasive Electrical Stimulation Acupuncture Points (NESAP)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
This was a small pilot study to determine safety of a TENS unit to deliver NESAP to newborn infants during routine heel sticks. The purpose was not to determine efficacy of NESAP to relieve pain during heel sticks. A large clinical trial will follow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes